CLINICAL TRIAL: NCT06925633
Title: The Impact of Supraphysiologic Estrogen Levels on Postoperative Recovery Quality in IVF Patients: A Prospective Observational Study
Brief Title: Estrogen Levels and Postoperative Recovery in IVF Patients
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 2.11.2024-33440
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: In Vitro Fertilization; Postoperative Recovery; Estrogens; Anesthesia Recovery Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate the relationship between supraphysiologic serum estrogen levels and postoperative recovery quality in patients undergoing IVF procedures under general anesthesia. Estrogen is known to play a role in pain modulation and emotional responses, both of which influence postoperative recovery. The primary outcome is the quality of recovery score (QoR-15), and secondary outcomes include postoperative pain, nausea and vomiting, and discharge time. A total of 100 adult female patients will be included. The study seeks to provide better insight into how elevated estrogen levels may impact patient outcomes after anesthesia.

DETAILED DESCRIPTION:
Postoperative recovery is a multidimensional and complex process influenced by pain, nausea and vomiting, emotional and functional factors. IVF (In Vitro Fertilization) treatments involve controlled ovarian hyperstimulation, which causes supraphysiologic increases in serum estrogen levels. Elevated estrogen is thought to affect pain modulation and inflammatory pathways and has been associated with increased symptoms such as nausea and mood fluctuations.

This prospective observational study aims to investigate the relationship between serum estrogen concentration and the quality of recovery in patients undergoing IVF-related transvaginal oocyte retrieval under general anesthesia. A total of 100 ASA I-II adult female patients between the ages of 18 and 45 will be enrolled.

Patients will be grouped based on their estradiol (E2) levels measured as part of the routine IVF procedure. E2 levels above 350 pg/ml will be defined as supraphysiologic. The primary outcome is the postoperative recovery quality assessed using the QoR-15 questionnaire at 24 and 72 hours postoperatively. Secondary outcomes include postoperative pain intensity (measured by the Numerical Rating Scale), nausea and vomiting (assessed by Verbal Descriptive Scale), and time to discharge (evaluated using the Modified Aldrete Score). Preoperative anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS).

This study aims to contribute to improved anesthetic and perioperative management of IVF patients with elevated estrogen levels.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 45 years
* ASA physical status I or II
* Scheduled for transvaginal oocyte retrieval under general anesthesia as part of an IVF procedure
* Willing and able to provide written informed consent
* Able to understand and complete study questionnaires (QoR-15, HADS)

Exclusion Criteria:

* ASA physical status III or IV
* History of severe renal, hepatic, respiratory, or cardiovascular disease
* Current or chronic use of psychotropic medications
* Chronic use of opioids or benzodiazepines
* Known psychiatric or neurological disorders that may interfere with study participation
* Inability to provide informed consent or complete study questionnaires

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: The study population consists of adult female patients aged 18 to 45 years undergoing transvaginal oocyte retrieval under general anesthesia as part of an IVF procedure. All participants will have ASA physical status I or II and be able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Recovery Quality (QoR-15 Score) | 24 hours and 72 hours after surgery
  Assessed using the Quality of Recovery-15 (QoR-15) questionnaire at 24 and 72 hours postoperatively. The score ranges from 0 to 150, with higher scores indicating better recovery.

SECONDARY OUTCOMES:
Postoperative Pain Intensity (NRS Score) | 24 and 72 hours after surgery
  Assessed using the Numerical Rating Scale (NRS) where 0 indicates no pain and 10 indicates worst imaginable pain.
Postoperative Nausea and Vomiting (VDS Score) | 24 and 72 hours after surgery
  Evaluated using the Verbal Descriptive Scale (VDS); scale ranges from 0 (none) to 4 (severe nausea and vomiting).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.